CLINICAL TRIAL: NCT03942666
Title: A Clinical Pharmacology Study to Evaluate the CHF 6532 Linearity After Single Oral Administrations of Four Doses of a Tablet Formulation Followed by an Evaluation of the Pharmacokinetic at Steady State Following the Repeated Open Label b.i.d. Administration at One Dose
Brief Title: PK Linearity and Steady State PK of CHF 6532 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: CLI-06532AA1-03; 2019-000250-59 (EudraCT Number)
Record Dates: First submitted 2019-05-06; First posted 2019-05-08 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Intervention Model Description: Part I: 5-way, 5-period crossover Part II: single group
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Part II: double blind Part II: open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Treatment A (Experimental): Single administration of CHF 6532 Dose #1
  Interventions: Drug: Treatment A
- Treatment B (Experimental): Single administration of CHF 6532 Dose #2
  Interventions: Drug: Treatment B
- Treatment C (Experimental): Single administration of CHF 6532 Dose #3
  Interventions: Drug: Treatment C
- Treatment D (Experimental): Single administration of CHF 6532 Dose #4
  Interventions: Drug: Treatment D
- Treatment E (Placebo Comparator): Single administration of CHF 6532 Placebo
  Interventions: Drug: Treatment E
- Treatment F (Other): Part II: Administration of tablet of CHF 6532 b.i.d. for 10 days at one dose.
  Interventions: Drug: Treatment F

INTERVENTIONS:
Drug: Treatment A — tablet of CHF 6532
  Arms: Treatment A
Drug: Treatment B — tablet of CHF 6532
  Arms: Treatment B
Drug: Treatment C — tablet of CHF 6532
  Arms: Treatment C
Drug: Treatment D — tablet of CHF 6532
  Arms: Treatment D
Drug: Treatment E — Placebo tablet of CHF 6532
  Arms: Treatment E
Drug: Treatment F — tablet of CHF 6532
  Arms: Treatment F

SUMMARY:
The purpose of this clinical pharmacology study is to evaluate the CHF 6532 linearity after single oral administrations of four doses of a tablet formulation and to evaluate the pharmacokinetic (PK) at steady state following the repeated open label b.i.d. administration at one dose.

DETAILED DESCRIPTION:
The study consists in two parts. The first study part (Part I) is a single dose, randomised, double-blind, placebo-controlled, 5-way, 5-period crossover design, in healthy subjects.

The second study part (Part II) is a repeated dose, open label treatment in healthy subjects.

The PK of CHF 6532 and CHF 6532 acyl glucuronide metabolite (CHF 6532-AG), the cardiac safety will be assessed after single or repeated administration of CHF 6532 tablet formulations in healthy subjects under fed conditions.

A total of 30 healthy male and female are planned to be included where they will participate the 2 study parts.

Standard safety assessments will be conducted during the Study, including safety blood and urine laboratory tests, vital signs, physical examinations, ECGs and observations of any adverse events. Blood and urines samples will be also collected for PK analysis. Holter recordings will be performed to build a prospective concentration-response model of QTc for CHF 6532 in Part I and for cardiac safety purpose at steady state in Part II.

ELIGIBILITY:
Inclusion Criteria:

* Subject's written informed consent obtained prior to any study-related procedure;
* Healthy male or female subjects aged 18-60 years inclusive;
* Ability to understand the study procedures, the risks involved and willingness to follow the study procedures including intake of non-permitted concomitant medications;
* Body Mass Index (BMI) between 19.0 and 30.0 kg/m2 extremes inclusive;
* Non- or ex-smokers who smoked < 5 pack years;
* Good physical and mental status, determined on the basis of the medical history and a general physical examination;
* Vital signs within normal limits;
* Body temperature 35.5-37.2ºC;
* 12-lead digitised Electrocardiogram (12-lead ECG) considered as normal;
* Female subject of non-childbearing potential (WONCBP) defined as physiologically incapable of becoming pregnant (i.e. post-menopausal or permanently sterile) and female subjects of childbearing potential (WOCBP) fulfilling one of the following criteria: a/ WOCBP with fertile male partners: they and/or their partner must be willing to use a highly effective birth control method from the signature of the informed consent and until the follow-up visit or b/WOCBP with non-fertile male partners: (contraception is not required in this case).

Exclusion Criteria:

* Clinically significant abnormal 24 hours Holter ECG at screening;
* Subjects with history of sustained and non-sustained cardiac arrhythmias (ECG demonstrated) and subjects with a family history of sudden cardiac death;
* Blood donation or blood loss (equal or more than 450 ml) less than 8 weeks prior to randomisation;
* Abnormal haemoglobin level;
* Subjects with history of asthma, including childhood asthma, COPD or any other chronic pulmonary diseases or condition;
* Positive HIV1 or HIV2 serology;
* Positive results for the Hepatitis serology;
* Clinically relevant and uncontrolled hepatic, gastrointestinal, endocrine, metabolic (specially, subjects with deficiency in glucuronidation), neurologic, or psychiatric disorder that may interfere with successful completion of this protocol according to the Investigator's judgement;
* Any clinically relevant abnormal laboratory value suggesting an unknown disease and requiring further clinical investigation or which may impact the safety of the subject or the evaluation of the result of the study according to the Investigator's judgment;
* Abnormal liver enzymes;
* Unsuitable veins for repeated venepuncture;
* History of substance abuse or drug abuse within 12 months prior to screening;
* Subjects who have received an investigational drug or device within 1 month or 7 times the elimination half-life (whichever is longer) prior to screening visit or are currently participating in another clinical trial or have been previously randomised in this trial;
* History of hypersensitivity to any of the excipients contained in the formulation used in the trial;
* Known intolerance/hypersensitivity to quinolone-type antibiotics, e.g. moxifloxacin, norfloxacin, ciprofloxacin, nalidixic acid;
* Heavy caffeine drinker;
* Subjects who have a positive urine test;
* Subject taking any drug treatment, including prescribed or OTC medicines as well as vitamins, homeopathic remedies etc, in the 14 days before the screening until randomisation, with the exception of: Occasional paracetamol, Hormonal contraceptives, Hormonal replacement treatment for post-menopausal women;
* Subject taking enzyme-inducing drugs, enzyme-inhibiting drugs, biologic drugs or any drug known to have a well-defined potential for hepatotoxicity (e.g. isoniazide, nimesulide, ketoconazole) in the 3 months before screening until randomisation;
* Pregnant or lactating women;
* History of risk factors for torsades de pointes, including unexplained syncope, known long QT syndrome, heart failure, myocardial infarction, angina or symptomatic arrhythmias. Subjects will also be excluded if there is a family history of long QT syndrome or Brugada syndrome or unexplained sudden death;
* Use of medications which are known to carry a risk of prolong the QTc interval is not allowed within 14 days or 7 times the elimination half-life (whichever is longer) before the baseline ECG.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-05-10 (Actual); Primary Completion 2019-11-22 (Actual); Study Completion 2019-11-22 (Actual)

PRIMARY OUTCOMES:
PK linearity of CHF 6532 | Over 12 hours after administration in urine, over 48 hours after administration in blood
  Assessment of CHF 6532 PK linearity in blood and urine depending on increasing doses of CHF 6532
Steady state PK of CHF 6532 | Over 12 hours after administration at Day 1 and Day 10 in urine, over 12 hours after administration at Day 1 and over 24 hours after administration at Day 10 in blood
  Assessment of CHF 6532 PK in blood and urine after a repeated administration of CHF 6532

SECONDARY OUTCOMES:
Cardiac Safety of CHF 6532 | Over 24 hours after single administration in Part I, Over 24 hours at Day 10 in Part II
  Holter recording
PK linearity of CHF 6532-AG | Over 12 hours after administration in urine, over 48 hours after administration in blood
  Assessment of CHF 6532-AG PK in blood and urine depending on increasing doses of CHF 6532
Steady state PK of CHF 6532-AG | Over 12 hours after administration at Day 1 and Day 10 in urine, over 12 hours after administration at Day 1 and over 24 hours after administration at Day 10 in blood
  Assessment of CHF 6532-AG PK in blood and urine after a repeated administration of CHF 6532

CONTACTS AND LOCATIONS:
Locations (1):
- SGS Life Sciences - Clinical Pharmacology Unit Antwerpen, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: No